CLINICAL TRIAL: NCT01145261
Title: The Relationship Between Emotional Regulation Strategies And Cognitive Behavioral Treatment Effectiveness In Childhood Anxiety Disorders: A Longitudinal Prospective Study
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, alan apter, Director Department of Psychological Medicine Schneider Children's Medical Center of Israel, Rabin Medical Center
Other Study IDs: 5846
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Anxiety
Keywords: Anxiety,; Emotional Regulation
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Anxiety: Children with anxiety disorders
- healthy controls: children without anxiety disorders

SUMMARY:
The current study will focus on two phases of anxiety process: Generating Anxiety (reported, direct and physiological) and Emotional Regulation Strategies (Reappraisal, Mindfulness, Expressive Suppression and Rumination). The claim is that better understanding of these phases in relation to CBT treatment will lead to better understanding of remission in anxiety and to better treatments in the future. Objectives: To understand the relations between the four strategies of emotional regulation to anxiety disorder hence to understand the relation between these strategies to treatment effectiveness of children with anxiety disorder. Methods: In phase one, clinically anxious adolescence before treatment (N=40) and healthy controls (N=40) will be compared. Anxious adolescence are expected to have significantly higher levels of physical arousal and will use spontaneously more expressive suppression and rumination and less reappraisal and mindfulness then the healthy controls. In phase two, clinically anxious adolescence (N=40) before and after 8-12 weeks of CBT treatment will be compared. More specifically remitted patients will be compared with partially remitted patients. Remitted patients are expected to show better improvement in the physical arousal, then partially remitted. More, Decrease in levels of anxiety will be mediated by the four emotional regulation strategies, and the efficiency of using the Reappraisal will be higher.

ELIGIBILITY:
Inclusion Criteria:

* anxious group: Clinical diagnosis of one or more of the following diagnoses: Generalized Anxiety Disorder, Social Anxiety, Separation Anxiety, panic disorder.
* non anxious group: do not meet the criteria for anxiety disorders as well as for any other mental disorder

Exclusion Criteria:

* anxious group: not treated during the study in any other treatment for anxiety disorders.Clinical diagnosis of one or more of the following diagnoses: psychosis, dyslexia, mental retardation, PTSD.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The anxious group: children who will present to the Anxiety Disorder Outpatient Clinic at Schneider Children's Hospital in Israel.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
level of anxiety - by cgi and scared scales | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Apter, MD, Principal Investigator — Director Department of Psychological Medicine Schneider Children's Medical Center of Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Departemnt of Psychological Medicine, Petah Tikva, Israel, Israel